CLINICAL TRIAL: NCT00135811
Title: Focal Segmental Glomerulosclerosis Clinical Trial
Brief Title: Focal Segmental Glomerulosclerosis Clinical Trial (FSGS-CT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Marva Moxey-Mims, M.D., NIH Project Officer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 63490 (completed)
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Glomerulosclerosis, Focal
Keywords: Focal Segmental Glomerulosclerosis
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental | interventions — Cyclosporine; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Cyclosporin
  Interventions: Drug: Cyclosporin
- 2 (Active Comparator): MMF and Dexamethasone
  Interventions: Drug: MMF and Dexamethasone

INTERVENTIONS:
Drug: Cyclosporin — Participants assigned to this group will initiate treatment with CSA, 5-6 mg/kg per day with a 250 mg/day maximum starting dose, divided into two daily doses. The CSA dose will be adjusted based on drug levels determined at specified study visits in order to achieve a 12-hour trough concentration in the therapeutic range of 100-250 ng/ml.
  Arms: 1
Drug: MMF and Dexamethasone — MMF, 25-36 mg/kg per day with a maximum dose of 2 g/day divided into two daily doses. The dose range reflects the use of fixed size (250 mg) capsules and application of defined daily doses to specific weight ranges (see Table below). In younger children or those participants who are unable to swallow capsules, a liquid formulation will be used to provide 36 mg/kg per day to a maximum of 2 g per day. The starting MMF dose will be 0.5-0.67 of the full dose for 2 weeks before advancing to the full dose for the duration of the 12-month treatment period.
  Dexamethasone, 0.9 mg/kg per dose, with a maximum dose of 40 mg
  Arms: 2

SUMMARY:
The FSGS Clinical Trial is a multi-center, prospective, controlled, open label randomized trial designed to determine if treatment with mycophenolate mofetil (MMF) in conjunction with pulse steroids is superior to treatment with Cyclosporine-A (CSA) in inducing remission from proteinuria over 12 months.

DETAILED DESCRIPTION:
Background/Rationale. Primary FSGS is a leading cause of end stage renal disease in both children and adults, with complete loss of kidney function in 50% of patients over 10 years. Evidence-based treatment guidelines for FSGS have not been developed because of the lack of controlled studies and the small number of patients included in most reports. Over the past decade, a number of studies have reported therapeutic efficacy for treatment with Cyclosporine-A (CSA) in patients with nephrotic syndrome including patients with steroid resistant FSGS. There have been two controlled trials of treatment with CSA in steroid resistant FSGS, one in children and one in adult patients. Consequently, CSA is the only medication that has been documented to be efficacious in a controlled trial in both children and adults with steroid resistant FSGS. The experience with mycophenolate mofetil (MMF) in the treatment of patients with steroid resistant FSGS has been limited to uncontrolled trials in adult patients and children.

Patient Population. The patient population consists of children and adults between the ages of 2 and 40 years with steroid resistant FSGS.

Study Design. The experimental design is a multi-center, prospective, controlled, open label randomized trial comparing two treatment regimens, CSA vs. MMF/Pulse Steroids. The treatment regimens in both arms also include angiotensin converting enzyme inhibitor (ACEI) therapy and alternate day low dose prednisone. The CSA and MMF/Pulse steroid treatment regimens will be implemented over the first 26 weeks after randomization and continued to 52 weeks if a response in proteinuria occurs. The ACE inhibitor component continues for an additional 26 weeks after withdrawal of initial therapies.

Logistical Structure. Participants are recruited at over 130 participating sites in North America which are affiliated with one of five Core Coordinating Centers.

Primary Objectives. The primary objective of the trial is to determine if treatment with MMF/Pulse steroids is superior to treatment with CSA in inducing remission from proteinuria over 12 months. The main secondary objective is to determine if treatment with MMF/Pulse steroids is superior to treatment with CSA in inducing remissions which persist for at least 6 months following withdrawal of immunosuppressive therapy but while maintaining ACEI or angiotensin receptor blocker (ARB) therapy.

Biorepository Specimens. Collection of specimens for biological and DNA repositories will serve as a national resource for ancillary studies investigating the pathogenesis of FSGS.

Duration of Therapeutic Regimens and Follow-up. The study treatment duration for a randomized patient depends on the level of response to treatment as follows: 26 weeks if neither a partial or complete remission occurs at the 26-week visit; 52 weeks if there is a partial or complete remission at 26 weeks but not at 52 weeks, and 78 weeks if partial or complete remissions are recorded at both the 26- and 52-week visits. For all patients low intensity follow-up for long-term assessment of renal function is maintained after termination of the therapeutic regimens until September, 2008.

Inclusion Criteria.

* Age 2-40 years at onset of signs or symptoms of FSGS,
* Age ≤ 40 years at randomization,
* Estimated glomerular filtration rate (GFR) ≥ 40 ml/min/1.73 m2,
* Urine protein/creatinine (Up/c) > 1.0 on first am void,
* Biopsy confirmed primary FSGS (including all subtypes),
* Steroid resistance established by failure to achieve a sustained Up/c < 1.0 following a steroid treatment course of at least 4 weeks with a minimum cumulative dose of 56 mg/kg or 1,680 mg of prednisone, and
* Willingness to follow the clinical trial protocol, including medications, and baseline and follow-up visits and procedures.

Exclusion Criteria.

* Secondary FSGS,
* Prior therapy with sirolimus, CSA, tacrolimus, MMF, or azathioprin (Imuran), - - Treated with cytoxan, chlorambucil, levamisole, methotrexate, or nitrogen mustard in the last 30 days,
* Lactation, pregnancy, or refusal of birth control in women of child bearing potential,
* Participation in another therapeutic trial concurrently or 30 days prior to randomization,
* Active/serious infection,
* Malignancy,
* Blood pressure > 140/95 or > 95th percentile for age/height,
* Use of 4 or more antihypertensive agents for the primary purpose of controlling blood pressure,
* Previously diagnosed diabetes mellitus type I or II (DM I or II),
* Clinical evidence of cirrhosis or chronic active liver disease,
* Absolute neutrophil count (ANC) < 2000/mm3 or hematocrit (HCT) < 28%,
* History of significant gastrointestinal disorder,
* Organ transplantation,
* Obesity (based on estimated dry weight at onset of disease prior to steroid therapy) defined as body mass index (BMI) > 97th percentile for ages 2-20 years, and BMI > 40 kg/m2 for age ≥21 years,
* Allergy to study medications, and 17) Inability to consent/assent.

Therapeutic Regimens.

CSA Arm:

CSA: The initial target dose for CSA is 5 - 6 mg/kg per day divided into two daily doses. Dosage is subsequently adjusted to maintain a 12-hour trough CSA blood concentration of 100 - 250 ng/ml. CSA is maintained for 12 months following randomization.

MMF/Pulse Steroid Arm:

MMF: The target dose for MMF is 25-36 mg/kg per day with a maximum dose of 2 g/day divided into two daily doses, maintained for 12 months following randomization.

Dexamethasone: The target dose for dexamethasone is 0.9 mg/kg per dose, with a maximum dose of 40 mg, given as a single dose on two consecutive days at the start of weeks 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 30, 34, 38, 42, 46 and 50 for a total of 46 doses.

Both Treatment Arms:

ACEI: A maximally tolerated dose of the angiotensin converting enzyme inhibitor, lisinopril will be attempted in three steps at two-week intervals. The target maintenance dose ranges from 0.4 mg/kg to 0.6 mg/kg depending on the patient's weight. Patients who are unable to tolerate treatment with ACEI or who have been previously intolerant of ACEI will receive the angiotensin receptor blocker (ARB) losartan. The duration for the ACEI or ARB therapy is 18 months.

Prednisone: Target dose for prednisone is 0.3 mg/kg per dose to a maximum dose of 15 mg, administered as single dose every other day for the first 6 months of the 12-month treatment period after randomization.

Dose Adjustments for Toxicity:

Known toxicities associated with each of the therapeutic agents are delineated in the protocol. A stepped dosage reduction protocol is implemented following confirmed toxicities as follows:

* Step 1: Reduce dosage to 2/3 of full target dose;
* Step 2: If the toxicity persists following Step 1, reduce dose to 1/3 of full target dose;
* Step 3: If the toxicity persists following Step 2, discontinue medication. In certain cases, the protocol stipulates that the attempts should be made to reverse the dose reductions (following the stepped sequence in reverse order) following remission of toxicities.

Study Visits and Measurements. Main Outcome Assessment Visits: The main visits for assessment of study outcomes are conducted at baseline and at weeks 26, 52, and 78 of follow-up. These visits each include 2 first-morning Up/c, a full panel of serum and urine biochemistry measurements, complete blood count, a quality of life assessment (SF-36 in adults; PedsQL in children), a complete physical examination, recording of medications and side effects, plus additional urine, serum, plasma specimens for storage in a repository. Whole blood for DNA extraction will be collected at onset of therapy and placed in a repository for consenting patients.

Other Visits: In addition to the main outcome assessment visits at baseline and weeks 26, 52, and 78, first morning urine samples for determination of Up/c, basic blood chemistries (BUN, creatinine, serum electrolytes and glucose) and hematology in the MMF/Pulse Steroids arm are also obtained immediately after randomization, and at follow-up weeks 2, 4, 6, 8, 14, 20, 32, 38, 44, and 65. CSA trough level, fasting lipids, serum albumin, and other blood chemistries are obtained at designated subsets of these visits.

Adverse event monitoring. Adverse events, including all hospitalizations, and all modifications to the dosages of the study medications are recorded throughout the follow-up period.

Definition of Partial and Complete Remissions. At each protocol assessment of proteinuria, a partial remission is defined as a 50% or greater decline in the first morning Up/c from the mean of two baseline measurements to a level between 0.2 and 1.0. A complete remission is defined as a decline in Up/c to a level no greater than 0.2.

Primary Outcome. The primary outcome is a 6-level ordinal classification based on the achievement of remission during the first 52 weeks after randomization. The least favorable outcome, designated as level 6, is assigned if no partial or complete remission is achieved between weeks 2 through 26, inclusive. Level 5 is assigned if the participant achieves at least one partial or complete remission between weeks 2 and 20, but does not achieve either a partial or complete remission at week 26. By this definition, the primary outcome is not affected by the Up/c after 26 weeks if a partial or complete remission is not achieved at 26 weeks, allowing those participants to switch to alternative therapies without affecting the primary analysis.

For participants with a partial or complete remission at week 26, a score between 1 and 4 is assigned depending on the remission status between week 26 and week 52. Level 4 is assigned if the participant fails to achieve either a partial or complete remission at week 52 or has a sustained relapse between weeks 26 and 52. Level 3 is assigned if the participant achieves a partial remission at week 52. Level 2 is assigned if the participant achieves a complete remission at week 52 but has had at least one Up/c > 0.2 after week 26 but before week 52. Level 1 is assigned if the participant achieves a complete remission at week 52 and has had Up/c < 0.2 since the week 26 visit.

Main Secondary Outcome. The main secondary outcome is a 5-level ordinal classification which evaluates the extent to which remissions from proteinuria persist during the period from week 52 to week 78 after immunosuppressive therapy is withdrawn but while remaining on ACEI or ARB treatment

Other Outcomes. Other outcomes include the change in quality of life, the numbers of adverse events and extra-renal complications, and preservation of renal function.

Sample Size. The target sample size is 500 patients.

Primary Analysis. The primary statistical analysis will compare the six-level primary outcome variable between the randomized treatment groups. The six levels will be assigned scores ranging from 1 (for the most favorable category) to 6 (for the least favorable category), and the mean response score will be compared between the CSA and MMF/Pulse steroid groups within each of the four randomization strata defined by baseline estimated GFR and race. The analysis will be carried out by intent-to-treat. A 2-sided test will be conducted at the 5% significance level.

Study Power. Depending on the remission rate in the control group (classified as levels 1, 2, or 3 for the primary outcome), the sample size of 500 randomized patients is sufficient to obtain 80% power to detect an absolute increase in remission rate of between 10.8% and 11.5% between the MMF/Pulse Steroid and the CSA groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-40 years at onset of signs or symptoms of FSGS
* Age ≤ 40 years at time of randomization (randomization date before 41st birthday)
* Estimated GFR ≥ 40 ml/min/1.73 m2 at most recent measure prior to randomization

  * For participants < age 18 years: Schwartz formula
  * For participants ≥ age 18 years: Cockroft-Gault formula
* Up/c > 1.0 g protein/g creatinine on first am void at time of randomization
* Biopsy confirmed as primary FSGS (including all subtypes) by study pathologist. A minimum of 1 glomerulus demonstrating segmental sclerosis on light microscopy will be required to confirm the diagnosis.
* Steroid resistance: The participant must have demonstrated steroid resistance (defined as a failure to achieve a sustained Up/c ≤ 1.0) based on at least one treatment course with high dose steroids prior to randomization which satisfies both of the following conditions:

  * minimal treatment duration of 4 weeks
  * minimum cumulative dose of 56 mg/kg or 1680 mg of prednisone or its equivalent. In addition, the participant must not have had a complete remission of proteinuria (Up/c < 0.2 or dipstick urine protein 0/trace) subsequent to the latest qualifying 4-week course demonstrating steroid resistance.
* Willingness to follow the clinical trial protocol, including medications, and baseline and follow-up visits and procedures.
* Participants may be taking ACEI, ARB, Vitamin E, or lipid lowering therapy.

Exclusion Criteria:

* Secondary FSGS
* Prior therapy with sirolimus, CSA, tacrolimus, MMF, or azathioprin (Imuran)
* Treated with cytoxan, chlorambucil, levamisole, methotrexate, or nitrogen mustard in the last 30 days
* Lactation, pregnancy, or refusal of birth control in women of child bearing potential
* Participation in another therapeutic trial concurrently or 30 days prior to randomization
* Active/serious infection (including, but not limited to Hepatitis B, C, or HIV)
* Malignancy
* Blood pressure > 140/95 or > 95th percentile for age/height.
* Participant is receiving 4 or more antihypertensive agents for the primary purpose of controlling blood pressure.
* Participants with previously diagnosed diabetes mellitus type I or II: the diagnosis of DM I or II will be based on local criteria for participants with an established diagnosis. If hyperglycemia is detected during the screening period, the WHO criteria for the diagnosis of DM I and II will be used.
* Clinical evidence of cirrhosis or chronic active liver disease
* Abnormal laboratory values at the time of study entry:

  * Absolute neutrophil count (ANC) < 2000/mm3, or
  * Hematocrit (HCT) < 28%
* History of significant gastrointestinal disorder, e.g, severe chronic diarrhea (> 5 watery stools per day) or active peptic ulcer disease.
* Organ transplantation
* Obesity (based on estimated dry weight at onset of disease prior to steroid therapy) defined as

  * BMI > 97th percentile for age if aged 2-20 years
  * BMI > 40 kg/m2 for age ≥21 years
* Allergy to study medications
* Inability to consent/assent

Note: Participants with conditions meeting exclusion criteria at a particular evaluation for eligibility may be re-evaluated at a later time to determine if the conditions have changed so that all entry criteria are met. In particular, if blood pressure > 140/95 or > 95th percentile for age/height while the participant is on less than three antihypertensive agents, the participant may be re-evaluated for eligibility after adding other antihypertensive agents so long as the total number of agents does not exceed three.

Ages: 2 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 207 (Estimated)
Dates: Start 2004-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome is a 6-level ordinal variable defined based on the achievement of remission from proteinuria during the first 52 weeks after randomization. | first 52 weeks after randomization.

SECONDARY OUTCOMES:
The main secondary outcome is a 5-level ordinal variable defined based on the persistence of remissions after immunosuppressive agents are withdrawn. | based on the participant's level of proteinuria during the period from week 52 through week 78 following withdrawal of CSA or MMF/Pulse steroids

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Friedman, MD, Study Chair — University of Minnesota; Marva Moxey-Mims, MD, FAAP, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- Data Coordinating Center; Cleveland Clinic Foundation; Quantitative Health Sciences; 9500 Euclid Avenue, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Liu ID, Willis NS, Craig JC, Hodson EM. Interventions for idiopathic steroid-resistant nephrotic syndrome in children. Cochrane Database Syst Rev. 2025 May 8;5(5):CD003594. doi: 10.1002/14651858.CD003594.pub7. PMID 40337980
- [Derived] Hodson EM, Sinha A, Cooper TE. Interventions for focal segmental glomerulosclerosis in adults. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD003233. doi: 10.1002/14651858.CD003233.pub3. PMID 35224732
- [Derived] Li Q, Gulati A, Lemaire M, Nottoli T, Bale A, Tufro A. Rho-GTPase Activating Protein myosin MYO9A identified as a novel candidate gene for monogenic focal segmental glomerulosclerosis. Kidney Int. 2021 May;99(5):1102-1117. doi: 10.1016/j.kint.2020.12.022. Epub 2021 Jan 4. PMID 33412162
- [Derived] Gipson DS, Trachtman H, Kaskel FJ, Greene TH, Radeva MK, Gassman JJ, Moxey-Mims MM, Hogg RJ, Watkins SL, Fine RN, Hogan SL, Middleton JP, Vehaskari VM, Flynn PA, Powell LM, Vento SM, McMahan JL, Siegel N, D'Agati VD, Friedman AL. Clinical trial of focal segmental glomerulosclerosis in children and young adults. Kidney Int. 2011 Oct;80(8):868-78. doi: 10.1038/ki.2011.195. Epub 2011 Jul 6. PMID 21734640
- [Derived] Gipson DS, Trachtman H, Kaskel FJ, Radeva MK, Gassman J, Greene TH, Moxey-Mims MM, Hogg RJ, Watkins SL, Fine RN, Middleton JP, Vehaskari VM, Hogan SL, Vento S, Flynn PA, Powell LM, McMahan JL, Siegel N, Friedman AL. Clinical trials treating focal segmental glomerulosclerosis should measure patient quality of life. Kidney Int. 2011 Mar;79(6):678-685. doi: 10.1038/ki.2010.485. Epub 2010 Dec 22. PMID 21178977